CLINICAL TRIAL: NCT06616740
Title: Comparison of the Effects of Paratracheal Compression and Cricoid Compression on LMA ProSeal Placement: a Randomised Clinical Trial.
Brief Title: Effects of Paratracheal Compression and Cricoid Compression on LMA ProSeal Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, muhammet korkusuz, Principal Investigator, MD, Karaman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 04-2024/16
Record Dates: First submitted 2024-09-23; First posted 2024-09-27 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Airway Management
Keywords: Airway management; LMA; Cricoid pressure; Paratracheal pressure; Supraglottic airway device

STUDY DESIGN:
Intervention Model Description: There are two groups;
  1. Experimental Group: Group P; paratracheal compression will be applied during LMA ProSeal insertion.
  2. Sham Comparator: Group C; cricoid compression will be applied during LMA ProSeal insertion.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: patients, care providers, investigator and outcome assessors will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cricoid pressure group (Sham Comparator): Cricoid pressure will be applied during LMA ProSeal insertion.
  Interventions: Other: Cricoid pressure
- Paratracheal pressure group (Experimental): Paratracheal pressure will be applied during LMA ProSeal insertion.
  Interventions: Other: Paratracheal pressure

INTERVENTIONS:
Other: Cricoid pressure — Cricoid pressure will be applied during LMA ProSeal insertion.
  Arms: Cricoid pressure group
Other: Paratracheal pressure — Pratracheal pressure will be applied during LMA ProSeal insertion.
  Arms: Paratracheal pressure group

SUMMARY:
The aim of this study is to compare the effect of paratracheal and cricoid pressure on LMA ProSeal insertion, insertion time, insertion difficulty, and the rate of optimal positioning of the device after insertion.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19-70 years who are scheduled for general anaesthesia for whom LMA management would be appropriate.

Exclusion Criteria:

* with cervical spine disease
* expected difficult airway
* upper airway abnormalities
* body mass index (BMI) more than 35 kg/m2
* high risk of aspiration (hiatus hernia, gastro-oesophageal reflux disease and starvation)
* postoperative ventilator care
* surgeries requiring positions other than supine.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-10-24 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Duration of insertion | During intubation procedure
  The time required for placement will be defined as the time from receipt of the LMA ProSeal to detection of the square waveform on capnography and will be calculated by summing the time taken for each attempt.

SECONDARY OUTCOMES:
Sensation of resistance during inserting of LMA ProSeal | During intubation procedure
  Insertion of the LMA ProSeal will be assessed on a 4-point scale (1, no resistance; 2, moderate resistance; 3, severe resistance; and 4, impossible to insert the LMA ProSeal).
Anatomical location of the LMA ProSeal in the larynx and accuracy of insertion site. | 1 minutes after intubation
  It will be evaluated with a fibreoptic bronchoscope placed inside the tube section of the the LMA ProSeal. Accuracy will be recorded on a five-point scale (1, only the glottis is observed; 2, the posterior surface of the epiglottis and the glottis are observed; 3, the anterior part or tip of the epiglottis and >50% of the glottis are observed; 4, the folded down epiglottis and <50% of the glottis are observed; 5, the glottis is completely hidden by the folded down epiglottis)
Tidal volume and peak inspiratory pressure with or without each maneuver after LMA ProSeal insertion. | 2 minutes after intubation
  Tidal volume and peak inspiratory pressure with or without manoeuvre will be recorded with the same ventilator settings determined for all patients.
Oropharyngeal leak pressure | 5 minutes after induction of general anesthesia
  Oropharyngeal leak pressure will be assessed by closing the expiratory valve of the circle system to 40 cmH2o, with a fresh gas flow of 3 L/min and noting the airway pressure when equilibrium is reached or an audible air leak occurs.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammet Korkusuz, MD, Principal Investigator — Karamanoglu Mehmetbey University, School of Medicine
Locations (1):
- Karaman Taining and Research Hospital, Karaman, Turkey (Türkiye)